CLINICAL TRIAL: NCT04407559
Title: Impact of the Rheumatoid Factor on Serological Testing Performance for Covid-19 in Rheumatoid Arthritis Patients
Brief Title: COVID-SErology in Rheumatoid Arthritis (COVID-19)
Acronym: COVID-SERA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0330
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID-19; Rheumatoid Arthritis
MeSH Terms: conditions — COVID-19; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Frozen serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Groupe 1: Group 1: Rheumatoid arthritis seropositive for RF (+)
  Interventions: Other: Serological analyses to be lead on a pre-existing biobank
- Groupe 2: Group 2: Rheumatoid arthritis seronegative for RF (-)
  Interventions: Other: Serological analyses to be lead on a pre-existing biobank

INTERVENTIONS:
Other: Serological analyses to be lead on a pre-existing biobank — 3 immunoassays will be used according to the procedure described (Demey-2020; Tuaillon-2020) :
  * WuHan UNscience Biotechnology Co., Ltd (Chine). COVID-19 IgG/IgM Rapid Test Kit, (Wuhan, China), will be refered as UNscience
  * Chongqing iSIA BIO-Technology Co., Ltd (Chine). 2019-nCoV IgM/IgG Diagnostic Test Kit ; (Chongqing, China), will be refered as iSIA
  * Xiamen Biotime Biotechnology Co. Ldt (Chine). (SARS-CoV-2) IgM/IgG Rapid Qualitative Test Kit, will be refered as Biotime.

SUMMARY:
Due to the Covid-19 worldwide outbreak, fragile patients with immune diseases, notably rheumatoid arthritis (RA), have to be even more specifically and carefully followed-up. However, it has been shown that false postive serological results often occured while detecting antibodies directed against SARS-CoV-2 in patients with positive rheumatodoid factor (RF). The investigators propose here to investigated this issue. Therefore, the investigators will test three different immunoassays on this specific population. The investigators aim to establish these assays specificity and the levels of RF for which there is a risk of anti-SARS-CoV-2 false positivity and thus ensure a better follow-up of RA patients. The RF isotype will be analysed to determine whether there is a correlation and the impact of the presence of anti-CCP (citrullinated cyclic antipeptide antibodies) will be studied and assessed.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common inflammatory rheumatism, affecting 0.5% to 1% of the European population. Characterized by symmetrical and distal erosive polyarthritis, its diagnosis is based on the association of the clinical assessment combined with the presence of a chronic biological inflammatory syndrome and of citrullinated cyclic antipeptide antibodies (CCP) and / or of rheumatoid factor. From a prognostic point of view, some factors allow the risk prediction of the progression to structural damage (bone erosion), such as the positivity of the rheumatoid factor or anti-CCP antibodies, and require the rapid introduction of basic immunosuppressive therapy or biotherapy. In the context of the SARS-CoV-2 pandemic, responsible for the COVID-19 disease, the interest of a serological test is essential from an epidemiological point of view in order to follow the evolution of the pandemic, and to adapt the strategy of de-confinement of the general population or of patients at risk. However, RA patients receiving biotherapy present an increased risk of infection. In this context of de-confinement, a SARS-CoV-2 serological analysis, before initiating RA patients future treatment or in order to adapt their current treatment, would be useful.

Detection of antibodies directed against SARS-CoV-2 by various detection kits is currently under evaluation. To the lack of serological test kits on the French market is added the complexity of verifying the sensitivity and specificity of these tests. On the other hand, the immune response to SARS-CoV-2 is complex and still quite unknown. The concomitant presence of several isotypes IgA, IgM and IgG is frequently observed. Thus, the isotypic switching of Ig does not seem to take place correctly in this disease case, which randers the serodiagnostics even more complicated to implement. Detection of the less specific IgMs would therefore be essential, in the case of SARS-CoV-2. Rheumatoid factor (RF) is an immunoglobulin (Ig), more often of the M type, directed against the Fc fragment of IgG. This antibody, although not directly pathogenic, is very frequently present in RA patients (70 to 80%), without being specific for this pathology since it can be observed in other autoimmune, infectious or hematological diseases as well. The presence of RF IgM, all the more in high titers, is problematic while performing many serological or immunological assays since these high levels can be responsible for false positive results.

During previous SARS epidemics (SARS-CoV-1 or MERS-CoV), false positive results of serological tests were observed. When detecting anti-SARS-CoV-1 IgG or IgM in patients who had not contracted SARS, the use of an ELISA kit, with plates coated with a cell lysate of Vero-E6 cells infected with SARS-CoV-1, had been shown to induce a low number of false positive results in healthy controls (less than 5%). However, the number of false positive results in patients with autoimmune diseases was much higher, and varied accordingly with the pathology (between 10% and 58%), the largest number of false positive results being obtained in lupus patients. This phenomenon can be explained by the use of an immune test using unpurified cell lysates, which contain antigens against which the autoantibodies present in the patient serum could react, thus distorting the outcome of the test. Other causes of increase in the false positive results rate have been described when performing SARS-CoV-1 serologies, such as the presence of active neoplasia, or because of a previous infection with another coronavirus. Indeed, other coronaviruses, such as HCoV-OC43 and HCoV-229E, display a nucleocapsid close to the one of SARS-CoV-1 : this similarity can be the source of cross-reactivity. The same phenomenon was observed with the latest coronavirus: it was therefore suggested to rather use recombinant antigens of SARS-CoV-2 in immunoassays, such as ELISA for instance Given the similarity between SARS-CoV1 and SARS-CoV2, it is likely that the various elements causing false positive results during serological tests for SARS-CoV-1, in particular the presence of auto-antibodies including RF, could also cause false positive results when performing serological tests targeting SARS-CoV-2. A recent Chinese study showed that a moderate or high rate of RF was associated with a significant rate of false positive results when searching for anti-SARS-CoV-2 IgM with a ELISA kit, which plates were however coated with recombinant antigen. The authors therefore proposed to include a urea dissociation step into the ELISA protocol, which seemed to improve the specificity of the test, without altering its sensitivity.

It thus appears essential to assess the influence of RF, for its different isotypes (IgG, IgM, IgA), on various serological tests for SARS-CoV-2 available in France, in order to better assess these tests specificity.

The investigators propose to evaluate and compare 3 different serological tests available for the detection of specific SARS-CoV-2 IgG and IgM. The rate of false positive results obtained for each type of test will be evaluated on sera originated from patients with RA who have never been in contact with SARS-CoV-2, since these sera were withdrawn before July 2019. The relation between the incidence of SARS-Cov-2 serological assays false positive results and RF antibody levels could be estimated, as well as the characterization of RF.

ELIGIBILITY:
Inclusion criteria:

- Samples from a pre-July 2019 RA patient biobank to ensure true negativity of Covid -19 (patients over 18 years old)

Exclusion criteria:

- Patients who have traveled to China or Saudi Arabia and therefore may have encountered other coronaviruses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis (RA) Patients monitored at Montpellier University Hospital Patients having an available and frozen serum sample withdrawn before July 2019 Patients over 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the false positive results rate | 4 months
  Evaluate the false positive results rate when using each one of the three SARS-CoV-2 serology tests in patients with rheumatoid factor plasma levels, so as to define the specificity of these tests in this RA population. all serum samples will be tested by the 3 different immunoassays. The RF plasma levels have already been measured (routine exam) and are written in the patients files. The results will be analysed, the data proceeded and hopefully we will be able to answer the question.

SECONDARY OUTCOMES:
Characterize the RF isotype (IgG, IgM or IgA) associated | 4 months
  Characterize the RF isotype (IgG, IgM or IgA) associated with the false positivity of the test.all serum samples will be tested by the 3 different immunoassays. The RF isotype will be established using the routine method and the results of anti-CCP and RF plasma levels are already known and this information is available in the patients files. The results will be analysed, the data proceeded and hopefully we will be able to answer the questions
Determine the influence of RA on the false positivity rate in subjects | 4 months
  Determine the influence of RA on the false positivity rate in subjects with negative RF titer. All serum samples will be tested by the 3 different immunoassays. The RF isotype will be established using the routine method and the results of anti-CCP and RF plasma levels are already known and this information is available in the patients files. The results will be analysed, the data proceeded and hopefully we will be able to answer the questions
Assess the influence of the presence of anti-CCP on the false positivity of the SARS-CoV-2 test | 4 months
  Assess the influence of the presence of anti-CCP on the false positivity of the SARS-CoV-2 test : all serum samples will be tested by the 3 different immunoassays. The RF isotype will be established using the routine method and the results of anti-CCP and RF plasma levels are already known and this information is available in the patients files. The results will be analysed, the data proceeded and hopefully we will be able to answer the questions.
Assess the relation between the RF plasma levels and the false positivity of the SARS-CoV-2 test | 4 months
  Assess the relation between the RF plasma levels and the false positivity of the SARS-CoV-2 test : all serum samples will be tested by the 3 different immunoassays. The RF isotype will be established using the routine method and the results of anti-CCP and RF plasma levels are already known and this information is available in the patients files. The results will be analysed, the data proceeded and hopefully we will be able to answer the questions.

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna FERREIRA, MD, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC